CLINICAL TRIAL: NCT03412773
Title: A Randomized, Open-label, Multicenter Phase 3 Study to Compare the Efficacy and Safety of BGB-A317 Versus Sorafenib as First-Line Treatment in Patients With Unresectable Hepatocellular Carcinoma
Brief Title: A Study of Tislelizumab Versus Sorafenib in Participants With Unresectable Hepatocellular Carcinoma (HCC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-301; 2017-002423-19 (EudraCT Number); CTR20170882 (Registry Identifier: ChinaDrugTrials); JapicCTI-194569 (Registry Identifier: Japic); RATIONALE-301 (Other: BeiGene)
Record Dates: First submitted 2018-01-03; First posted 2018-01-26 (Actual); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Hepatocellular Carcinoma (HCC)
Keywords: Advanced liver cancer; RATIONALE-301
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab; Sorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Safety Run-In Sub-study (Experimental): Japanese participants received 200 mg intravenous tislelizumab every 3 weeks to assess preliminary safety and tolerability.
  Interventions: Drug: Tislelizumab
- Arm A: Tislelizumab (Experimental): Participants received 200 mg of intravenous tislelizumab every 3 weeks until intolerable toxicity, withdrawal of consent, or the investigator determined no further benefit from the therapy.
  Interventions: Drug: Tislelizumab
- Arm B: Sorafenib (Active Comparator): Participants received 400 mg of oral sorafenib twice daily until intolerable toxicity, consent withdrawal, or the investigator deemed no further benefit.
  Interventions: Drug: Sorafenib

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200 mg intravenously (IV) once every three weeks (Q3W)
  Other Names: BGB-A317
  Arms: Arm A: Tislelizumab; Safety Run-In Sub-study
Drug: Sorafenib — Sorafenib 400 mg orally (PO) twice daily (BID)
  Other Names: Nexavar; BAY43-9006
  Arms: Arm B: Sorafenib

SUMMARY:
This Phase 3 study was a global, multicenter trial that randomly assigned participants to either tislelizumab or sorafenib as a first-line treatment for adults with advanced liver cancer (hepatocellular carcinoma) that could not be surgically removed. Before enrolling Japanese participants in the main Phase 3 study, a preliminary assessment of safety and tolerability (the Safety Run-In Sub-study) was conducted in Japan.

ELIGIBILITY:
Safety Run-In Sub-study Eligibility Criteria: The study included adult Japanese participants (≥ 20 years) with histologically confirmed hepatocellular carcinoma (HCC) at Barcelona Clinic Liver Cancer (BCLC) Stage C or B. Eligible participants had either received, were ineligible for, or declined standard treatment. Additional requirements were a Child-Pugh A classification within 7 days before enrollment, at least one measurable lesion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1, and an Eastern Cooperative Oncology Group (ECOG) Performance Status score of ≤ 1.

Main Study Key Inclusion Criteria:

1. Histologically confirmed diagnosis of HCC
2. Barcelona Clinic Liver Cancer (BCLC) Stage B or C disease not amenable to or progressing after loco-regional therapy and not amenable to a curative treatment approach
3. No prior systemic therapy for HCC (with the exception of HCC participants enrolled in the safety run-in substudy [Japan only])
4. Measurable disease
5. Child-Pugh score A
6. Easter Cooperative Oncology Group (ECOG) Performance Status ≤ 1
7. Adequate organ function

Main Study Key Exclusion Criteria:

1. Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC histology
2. Tumor thrombus involving main trunk of portal vein or inferior vena cava
3. Loco-regional therapy to the liver within 28 days before randomization
4. Clinical evidence of portal hypertension with bleeding esophageal or gastric varices at Screening, or within 6 months before randomization
5. Bleeding or thrombotic disorder or any prescribed anticoagulant requiring therapeutic international normalized ratio monitoring (eg, warfarin or similar agents) at Screening, or within 6 months before randomization/enrollment
6. Presence at Screening of active immune deficiency or autoimmune disease and/or prior history of any immune deficiency or autoimmune disease that may relapse
7. Participant with any condition requiring systemic treatment with either corticosteroids (> 10 mg daily of prednisone or equivalent) or other immunosuppressive medication within 14 days before randomization
8. History of interstitial lung disease or non-infectious pneumonitis, unless induced by radiation therapy
9. QT interval corrected for heart rate (QTc) (corrected by Fridericia's method) > 450 msec at Screening

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2017-12-18 (Actual); Primary Completion 2022-07-11 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, MD, Study Director — BeiGene
Locations (122):
- United States (9):
  - Providence Medical Foundation, Fullerton, California
  - UCLA Hematologyoncology, Los Angeles, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Umdnj Njms, Newark, New Jersey
  - Rj Zuckerberg Cancer Center, Lake Success, New York
  - Xcancerdayton Physician Network, Dayton, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ut Health San Antonio Mays Cancer Center, San Antonio, Texas
- China (37):
  - The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Military Hospital of China, Beijing, Beijing Municipality
  - Beijing Youan Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chinese Pla General Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat Sen Memorial Hospital, Sun Yat Sen University (North), Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital, Sun Yat Sen University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University Wuhan, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - General Hospital of Eastern Theater Command, Nanjing, Jiangsu
  - Jiangsu Province Cancer Hospital, Nanjing, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Jilin Province Peoples Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an, Shaanxi
  - The Affiliated Hospital of Qingdao University Branch Laoshan, Qingdao, Shandong
  - Weifang Peoples Hospital, Weifang, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
- Czechia (2):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni Nemocnice V Motole, Prague
- France (13):
  - Chu Caen Normandie, Caen
  - Hopital Beaujon, Clichy
  - Chu Besancon Hopital Jean Minjoz, Doubs
  - Chu de Grenoble Oncology, Grenoble
  - Chru de Lille Hopital Claude Huriez Hepato Gastro Enterologie, Lille
  - Chu Montpellier Hopital Saint Eloi, Montpellier
  - Centre Hospitalier Universitaire Nantes Hotel Dieu, Nantes
  - Hopital Larchet Chu Nice, Nice
  - Chu de Poitiers Site de La Mileterie, Poitiers
  - Hopital Robert Debre, Reims
  - Chu Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Paul Brousse Aphp, Villejuif
  - Institut Gustave Roussy, Villejuif
- Germany (7):
  - Charite Universitatsmedizin Berlin, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Uniklinik Koln (Aor), Cologne
  - Universitatsklinikum Dusseldorf, Düsseldorf
  - Kliniken Essen Mitte Evang Huyssens Stiftung, Essen
  - Medizinische Hochschule Hannover, Hanover
  - Universitaetsklinikum Leipzig Aor, Leipzig
- Italy (7):
  - Policlinico Sorsola Malpighi, Aou Di Bologna, Bologna
  - Po Di Cremona, Asst Di Cremona Oncologia Medica, Cremona
  - Universita Degli Studi Di Modena Azienda Ospedaliere Policlinco, Modena
  - Irccs Policlinico San Matteo, Universita Degli Studi Di Pavi, Pavia
  - Ulssdolomiti, Peschiera del Garda
  - Po Umberto I, Ao Ordine Mauriziano, Torino
  - Osp Sbortolo, Ulss Berica, Vicenza
- Japan (26):
  - Fujita Health University Hospital, Toyoake, Aichi-ken
  - Ehime Prefectural Central Hospital Gastroenterologic Medicine, Matsuyama, Ehime
  - National Hospital Organization Kyushu Medical Center, Fukuokacity, Fukuoka
  - Ogaki Municipal Hospital Gastroenterological Medicine, Ōgaki, Gifu
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Medical University Hospital, Nishinomiyashi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Yahabacho Shiwagun, Iwate
  - Yokohama City University Medical Center Gastroenterological Center, Yokohama, Kanagawa
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - National Hospital Organization Nagasaki Medical Center Gastroenterology, Ōmura, Nagasaki
  - Nho Osaka National Hospital, Osakashi, Osaka
  - Osaka International Cancer Institute, Osakashi, Osaka
  - Kindai University Hospital, Sayama, Osaka
  - Osaka University Hospital, Suitashi, Osaka
  - Sasaki Foundation Kyoundo Hospital Hepatology, Bunkyoku, Tokyo
  - Nihon University Itabashi Hospital Gastroenterological Surgery, Itabashiku, Tokyo
  - Japanese Red Cross Medical Center Gastroenterology, Shibuyaku, Tokyo
  - Center Hospital of the National Center For Global Health and Medicine, Shinjukuku, Tokyo
  - Wakayama Medical University, Wakayama, Wakayama
  - Chiba University Hospital Gastroenterological Medicine, Chiba
  - Kumamoto University Hospital, Kumamoto
  - University Hospital, Kyoto Prefectural Univ of Medicine, Kyoto
  - Osaka City General Hospital, Osaka
  - Osaka Metropolitan University Hospital, Osaka
  - Tottori University Hospital Multidisciplinary Internal Medicine, Tottori
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Clinical Research Center Sp Z Oo, Medic R Sp K, Poznan
  - Narodowy Instytut Onkologii Im Marii Skodowskiej Curie Pastwowy Instytut Badawczy, Warsaw
  - Centrum Badan Klinicznych, Wroclaw
- Spain (4):
  - Hospital Universitario Vall Dhebron, Barcelona
  - Institut Catala Doncologia, Barcelona
  - Hospital Universitario Hm Madrid Sanchinarro, Madrid
  - Hospital Universitari I Politecnic La Fe, Valencia
- Taiwan (9):
  - Kaohsiung Medical University Chung Ho Memorial Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital Gastroenterology, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center, Tainan
  - Taipei Veterans General Hospital, Taipei
  - Tri Service General Hospital, Taipei
  - Linkou Chang Gung Memorial Hospital, Taoyuan District
- United Kingdom (4):
  - Queen Elizabeth Hospital, Birmingham
  - The Christie Hospital, Greater Manchester
  - Royal Free Hospital London Nhs Trust, London
  - Kings College, London

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Qin S, Finn RS, Kudo M, Meyer T, Vogel A, Ducreux M, Macarulla TM, Tomasello G, Boisserie F, Hou J, Li X, Song J, Zhu AX. RATIONALE 301 study: tislelizumab versus sorafenib as first-line treatment for unresectable hepatocellular carcinoma. Future Oncol. 2019 Jun;15(16):1811-1822. doi: 10.2217/fon-2019-0097. Epub 2019 Apr 10. PMID 30969136
- [Result] Qin S, Kudo M, Meyer T, Bai Y, Guo Y, Meng Z, Satoh T, Marino D, Assenat E, Li S, Chen Y, Boisserie F, Abdrashitov R, Finn RS, Vogel A, Zhu AX. Tislelizumab vs Sorafenib as First-Line Treatment for Unresectable Hepatocellular Carcinoma: A Phase 3 Randomized Clinical Trial. JAMA Oncol. 2023 Dec 1;9(12):1651-1659. doi: 10.1001/jamaoncol.2023.4003. PMID 37796513
- [Result] Finn RS, Kudo M, Barnes G, Meyer T, Boisserie F, Abdrashitov R, Chen Y, Li S, Zhu AX, Qin S, Vogel A. Tislelizumab versus Sorafenib in First-Line Treatment of Unresectable Hepatocellular Carcinoma: Impact on Health-Related Quality of Life in RATIONALE-301 Study. Liver Cancer. 2024 Feb 21;13(5):548-560. doi: 10.1159/000537966. eCollection 2024 Oct. PMID 39435268

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The main study enrolled participants across centers in Asia, Europe, and the U.S. The first participant consented on December 18, 2017, and the study concluded on December 14, 2023. In Japan, a safety run-in sub-study was conducted to evaluate tislelizumab's safety and tolerability in Japanese patients with hepatocellular carcinoma (HCC). Sub-study participants were not assessed for the same primary and secondary endpoints specified for the main study.
Pre-assignment Details: The main study had 4 phases: Screening, Treatment, Safety Follow-up (up to 30 days post-treatment or 90 days post-tislelizumab for immune events); and Survival Follow-up (duration varied). Randomization in the main study was stratified by macrovascular invasion (present vs absent), extrahepatic spread (present vs absent), etiology (hepatitis C virus vs other), Eastern Cooperative Oncology Group Performance Status (0 vs 1) and geography (Asia [excluding Japan] vs Japan vs Rest of World).
Period: Overall Study
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib
Started | 10 | 342 | 332
Treated | 10 | 338 | 324
Completed | 0 | 0 | 0
Not Completed | 10 | 342 | 332
Not completed — Lost to Follow-up | 0 | 7 | 6
Not completed — Withdrawal by Subject | 0 | 15 | 19
Not completed — Study Closed By Sponsor | 3 | 46 | 33
Not completed — Transfer to Long Term Extension (BGB-A317-290-LTE1) or Post Trial Supply (PTS) | 0 | 15 | 0
Not completed — Death | 7 | 259 | 273
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Sub-study: Safety Analysis Set includes all participants in the safety run-in sub-study who received at least one dose of any study drug.
  Main Study: Intent-to-Treat Analysis Set includes all participants randomized in the main study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib | Total
Number analyzed (Participants) | 10 | 342 | 332 | 684
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.70 (8.247) | 60.45 (12.528) | 59.51 (12.737) | 60.15 (12.652)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 53 | 51 | 107
  Male | 7 | 289 | 281 | 577
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 10 | 255 | 250 | 515
  White | 0 | 71 | 73 | 144
  Not Reported | 0 | 9 | 6 | 15
  Unknown | 0 | 4 | 1 | 5
  Black or African American | 0 | 3 | 2 | 5
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0
Eastern Cooperative Oncology Group (ECOG) Performance Status [Count of Participants; unit: Participants] — The ECOG scale assesses disease status from 0 to 5. A score of 0 means fully active with no restrictions, while 1 indicates limitations in strenuous activities but the ability to do light work. Score 2 signifies ambulatory and capable of self-care, yet unable to work, being active for over 50% of waking hours. Score 3 reflects limited self-care, confined to bed or a chair for more than half the day. Score 4 indicates complete disability, with the participant fully bedbound, and score 5 means deceased.
  Participants
    0 (Fully active) | 9 | 182 | 180 | 371
    1 (Restricted but ambulatory) | 1 | 160 | 152 | 313
Macrovascular Invasion [Count of Participants; unit: Participants] — Macrovascular invasion refers to the spread of cancer into large blood vessels near the tumor, and is associated with a more advanced stage of disease and a poorer prognosis. When present, cancer has infiltrated major blood vessels; when absent, no invasion into these vessels is detected, indicating a less aggressive disease.
  Participants
    Present | 0 | 51 | 48 | 99
    Absent | 10 | 291 | 284 | 585
Extrahepatic Spread [Count of Participants; unit: Participants] — Extrahepatic spread refers to the spread of liver cancer beyond the liver to other organs or tissues. When present, cancer has metastasized outside the liver; when absent, the cancer is confined to the liver.
  Participants
    Present | 4 | 219 | 198 | 421
    Absent | 6 | 123 | 134 | 263
Geographic Region [Number; unit: participants]
  Asia (excluding Japan) | 0 | 215 | 210 | 425
  Japan | 10 | 38 | 39 | 87
  European Union (EU)/United States (US) | 0 | 89 | 83 | 172
Etiology [Count of Participants; unit: Participants] — Participants were grouped based on the presence of Hepatitis C virus or another virus, with those having both Hepatitis B and C classified under the "other" category.
  Participants
    Hepatitis C Virus | 4 | 46 | 39 | 89
    Other | 6 | 296 | 293 | 595

OUTCOME MEASURES:

1. Primary Outcome: Safety Run-in Sub-study: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any unfavorable or unintended sign (e.g., abnormal lab result), symptom, or disease temporally associated with study drug use, regardless of causality.
  A serious adverse event (SAE) is defined as any adverse event that:
  * Resulted in death
  * Was life-threatening
  * Required or prolonged hospitalization
  * Caused disability/incapacity
  * Lead to a congenital anomaly/birth defect
  * Was deemed medically significant by the investigator (e.g., required intervention to prevent severe outcomes).
Time Frame: From the first dose to 30 days after the last dose, new anticancer therapy, or the analysis cutoff of December 14th, 2023 (a maximum of 64 months)
Population: The Sub-study Safety Analysis Set includes all participants in the safety run-in sub-study who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In Sub-study
Number analyzed (Participants) | 10
Participants
  TEAEs | 8
  SAEs | 1

2. Primary Outcome: Safety Run-in Sub-study: Serum Concentration of Tislelizumab
Description: Serum concentration of tislelizumab was a pre-specified primary endpoint for the sub-study only.
Time Frame: Cycle 1 and Cycle 5 at end of infusion, 24 hand 72 hours post-dose, and 8 days and 15 days post-dose (each cycle was 3 weeks).
Population: The Sub-study Pharmacokinetic (PK) Analysis Set includes all participants in the safety run-in sub-study who received at least 1 dose of tislelizumab per the protocol, for whom any post-dose PK data were available at each time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/mL
Arm/Group | Safety Run-In Sub-study
Number analyzed (Participants) | 10
µg/mL
  Cycle 1 End of Infusion | 63.21 (22.304)
  Cycle 1: 24 Hours Post Dose | 53.04 (20.901)
  Cycle 1: 72 Hours Post Dose | 42.06 (23.649)
  Cycle 1: 8 Days Post Dose | 32.61 (16.920)
  Cycle 1: 15 Days Post Dose | 23.74 (18.328)
  Cycle 5 Day 1: Predose: number analyzed (Participants) | 6
  Cycle 5 Day 1: Predose | 27.17 (34.436)
  Cycle 5 Day 1: End of Infusion: number analyzed (Participants) | 6
  Cycle 5 Day 1: End of Infusion | 87.54 (27.508)
  Cycle 5: 24 Hours Post Dose: number analyzed (Participants) | 6
  Cycle 5: 24 Hours Post Dose | 80.54 (27.006)
  Cycle 5: 72 Hours Post Dose: number analyzed (Participants) | 6
  Cycle 5: 72 Hours Post Dose | 64.80 (23.837)
  Cycle 5: 8 Days Post Dose: number analyzed (Participants) | 6
  Cycle 5: 8 Days Post Dose | 52.65 (26.759)
  Cycle 5: 15 Days Post Dose: number analyzed (Participants) | 6
  Cycle 5: 15 Days Post Dose | 37.57 (24.982)

3. Primary Outcome: Main Study: Overall Survival (OS)
Description: Defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using Kaplan-Meier methodology. Overall survival was a pre-specified primary endpoint for the main study only.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: The Intent-To-Treat (ITT) analysis set included all randomized participants in the main study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
Months | 15.9 [13.2 to 19.7] | 14.1 [12.6 to 17.4]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Non-Inferiority — Overall survival (OS) was compared between the tislelizumab group (Arm A) and the sorafenib group (Arm B) by testing the null hypothesis of noninferiority: the null hypothesis assumes the hazard ratio (HR) for tislelizumab versus sorafenib is greater than or equal to 1.08, while the alternative hypothesis assumes the hazard ratio is less than 1.08. Noninferiority was declared if the upper limit of the 95.003% confidence interval (CI) for the HR was less than 1.08; Hazard Ratio (HR) = 0.85, 95.003% CI 2-sided [0.712 to 1.019] — The hazard ratio is based on a Cox regression model with treatment, geography (Asia vs. EU/US), macrovascular invasion/extrahepatic spread (present vs. absent), etiology (HCV vs. other), and ECOG (0 vs. 1) as covariates
Statistical Analysis 2: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Superiority — Superiority of tislelizumab over sorafenib was tested for OS using a stratified log-rank test in the ITT analysis set only when noninferiority was demonstrated. Superiority was declared if the one-sided p-value crosses the boundary of 0.0223 (1-sided p-value < 0.0223) in favor of Arm A in the stratified log-rank test; p = 0.0398, Log Rank — One sided Log-Rank Test stratified by geography (Asia vs EU/US), macrovascular invasion and/or extrahepatic spread (present vs. absent), etiology (HCV vs. Other) and ECOG (0 vs. 1); Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.712 to 1.019] — The hazard ratio was derived from a Cox regression model with treatment as a covariate and stratified by geography (Asia vs. EU/US), macrovascular invasion/extrahepatic spread (present vs. absent), etiology (HCV vs. other), and ECOG score (0 vs. 1)

4. Secondary Outcome: Overall Response Rate (ORR) as Assessed by Blinded Independent Review Committee (BIRC)
Description: Defined as the percentage of participants who had partial response or complete response as determined by Blinded Independent Review Committee (BIRC) per the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 in all randomized participants with measurable disease at baseline.
  ORR was not assessed by the BIRC for participants in the sub-study, and this was not a pre-specified sub-study endpoint.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
percentage of participants | 14.3 [10.8 to 18.5] | 5.4 [3.2 to 8.4]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; The null hypothesis assumed that ORR is equal in both groups, while the alternative hypothesis assumed ORR is higher in the tislelizumab group (Arm A); Test type: Other; p = 0.0003, Cochran-Mantel-Haenszel — The nominal P-value from the Cochran-Mantel-Haenszel chi-square test, conducted at a 0.05 significance level, was stratified by geography, macrovascular invasion/extrahepatic spread, etiology, and ECOG; Cochran-Mantel-Haenszel ORR difference = 8.28, 95% CI 2-sided [3.85 to 12.70]

5. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator
Description: Defined as the percentage of participants who had partial response or complete response as determined by the investigator per RECIST v1.1 in all randomized participants with measurable disease at baseline.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: Sub-study Safety Analysis Set; Main study ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 10 | 342 | 332
percentage of participants | 20 [2.5 to 55.6] | 15.5 [11.8 to 19.8] | 5.7 [3.5 to 8.8]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 4, analysis 1]; Cochran-Mantel-Haenszel ORR difference = 9.24, 95% CI 2-sided [4.71 to 13.78]

6. Secondary Outcome: Progression Free Survival (PFS) as Assessed by BIRC
Description: Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as assessed by the BIRC per RECIST v1.1. Kaplan-Meier methodology was used to estimate the median PFS.
  PFS was not assessed by the BIRC for participants in the sub-study, and this was not a pre-specified sub-study endpoint.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
months | 2.1 [2.1 to 3.5] | 3.4 [2.2 to 4.1]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Other; p = 0.1364, One-sided log-rank test — [p-value comment as in outcome 3, analysis 2]; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.92 to 1.33] — [estimate comment as in outcome 3, analysis 2]

7. Secondary Outcome: Progression Free Survival (PFS) Assessed by the Investigator
Description: Defined as the time from randomization to the first objectively documented disease progression, or death from any cause, whichever occurred first, as assessed by the investigator per RECIST v1.1. Kaplan-Meier methodology was used to estimate the median PFS.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: Sub-study Safety Analysis Set; Main study ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 10 | 342 | 332
Months | 2.1 [1.9 to 16.0] | 2.1 [2.1 to 2.3] | 4.0 [2.7 to 4.1]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Other; p = 0.2622, One-sided log-rank test — [p-value comment as in outcome 3, analysis 2]; Hazard Ratio (HR) = 1.06, 95% CI 2-sided [0.90 to 1.26] — [estimate comment as in outcome 3, analysis 2]

8. Secondary Outcome: Duration of Response (DOR) as Assessed by BIRC
Description: Defined as the time from the first occurrence of a documented objective response until the first documentation of progression or death from any cause, whichever occurred first, as determined by the BIRC per RECIST v1.1. Median DOR was estimated using Kaplan-Meier methodology.
  DOR was not assessed by the BIRC for participants in the sub-study, and this was not a pre-specified sub-study endpoint.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in the analysis, and percentages were based on the number of responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 49 | 18
months | 36.1 [16.8 to NA] — Not estimable due to insufficient number of participants with events | 11.0 [6.2 to 14.7]

9. Secondary Outcome: Duration of Response (DOR) Assessed by the Investigator
Description: Defined as the time from the first occurrence of a documented objective response until the first documentation of progression or death from any cause, whichever occurred first, as assessed by the investigator per RECIST v1.1. Median DOR was estimated using Kaplan-Meier methodology.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: Sub-study Safety Analysis Set; Main study ITT Analysis Set; Only participants with best overall response of complete response or partial response per investigator assessment were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 2 | 53 | 19
Months | NA [NA to NA] — Not estimable due to insufficient number of participants with events | 25.2 [18.1 to 46.8] | 13.8 [6.2 to 20.3]

10. Secondary Outcome: Time to Progression (TTP) Assessed by BIRC
Description: Defined as the time from the date of randomization to the date of the first objectively documented tumor progression as assessed by the BIRC per RECIST v1.1. Median TTP was estimated using Kaplan-Meier methodology.
  TTP was not assessed by the BIRC for participants in the sub-study, and this was not a pre-specified sub-study endpoint.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
Months | 2.2 [2.1 to 3.6] | 4.1 [2.2 to 4.1]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Other; p = 0.0859, One-sided log-rank test — [p-value comment as in outcome 3, analysis 2]; Hazard Ratio (HR) = 1.14, 95% CI 2-sided [0.94 to 1.38] — [estimate comment as in outcome 3, analysis 2]

11. Secondary Outcome: Time to Progression (TTP) as Assessed by the Investigator
Description: Defined as the time from the date of randomization to the date of the first objectively documented tumor progression as assessed by the investigator per RECIST v1.1. Median TTP was estimated using Kaplan-Meier methodology.
  TTP was not a pre-specified sub-study endpoint.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
months | 2.1 [2.1 to 3.3] | 4.1 [3.4 to 4.2]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Test type: Other; p = 0.1182, One-sided log-rank test — [p-value comment as in outcome 3, analysis 2]; Hazard Ratio (HR) = 1.12, 95% CI 2-sided [0.94 to 1.34] — [estimate comment as in outcome 3, analysis 2]

12. Secondary Outcome: Safety Run-in Sub-study: Overall Survival
Description: Defined as the time from the date of randomization to the date of death due to any cause. Median OS was estimated using Kaplan-Meier methodology.
Time Frame: Up a to 64 months
Population: Sub-study Safety Analysis Set
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Safety Run-In Sub-study
Number analyzed (Participants) | 10
months | 29.7 [3.0 to NA] — Not estimable due to insufficient number of participants with events

13. Secondary Outcome: Disease Control Rate (DCR) as Assessed by BIRC
Description: Defined as the percentage of participants whose best overall response (BOR) was complete response, partial response, or stable disease as assessed by the BIRC per RECIST v1.1.
  DCR was not a pre-specified endpoint for participants in the sub-study.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
percentage of participants | 44.2 | 50.3

14. Secondary Outcome: Disease Control Rate (DCR) as Assessed by the Investigator
Description: Defined as the percentage of participants whose best overall response (BOR) was complete response, partial response, or stable disease as assessed by the investigator per RECIST v1.1.
  DCR was not a pre-specified endpoint for participants in the sub-study.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
percentage of participants | 44.2 | 52.4

15. Secondary Outcome: Clinical Benefit Rate (CBR) as Assessed by BIRC
Description: Defined as the percentage of participants whose best overall response (BOR) was complete response, partial response, or stable disease greater than or equal to 24 weeks in duration, as assessed by the BIRC per RECIST v1.1.
  CBR was not a pre-specified endpoint for participants in the sub-study.
Time Frame: Through the primary analysis data cut-off date of July 11th, 2022 (up to approximately 55 months)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
percentage of participants | 25.4 | 24.4

16. Secondary Outcome: Clinical Benefit Rate (CBR) as Assessed by the Investigator
Description: Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or stable disease greater than or equal to 24 weeks in duration, as assessed by the investigator per RECIST v1.1.
  CBR was not a pre-specified endpoint for participants in the sub-study.
Time Frame: Through the study completion data cut-off date of December 14th, 2023 (up to approximately 65 months)
Population: ITT Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 342 | 332
percentage of participants | 25.7 | 28.9

17. Secondary Outcome: Change From Baseline in the European Organisation for Research and Treatment of Cancer Quality of Life Questionnaire-Hepatocellular Carcinoma 18 Questions (EORTC QLQ HCC 18) Index Score at Cycle 4
Description: The EORTC QLQ-HCC18 is a questionnaire specifically designed to assess health-related quality of life in participants with hepatocellular carcinoma. It includes six symptom scales measuring Fatigue (3 items), Jaundice (2 items), Body Image (2 items), Nutrition (5 items), Pain (2 items), Fever (2 items) and two single items measuring Sex Life and Abdominal Swelling. Participants respond on a scale from 1 = "Not at all" to 4 = "Very Much. Raw scores are transformed into a 0 to 100 scale using linear transformation. The HCC18 Index score is calculated from each of the 6 symptom scales and the 2 single items, and ranges from 0 to 100. Higher scores indicate greater symptom burden or worse quality of life.
  The EORTC QLQ-HCC18 was not assessed for participants in the sub-study.
Time Frame: Baseline to Cycle 4 (each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both Baseline and Cycle 4 are included
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 220 | 176
score on a scale | 1.6 [0.4 to 2.9] | 3.9 [2.6 to 5.2]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; Between-arm differences in the change from Baseline were assessed using a mixed model for repeated measures. The model included Baseline scores, stratification factors, treatment arms, visits, and treatment arm by visit interaction as fixed effects and visit as a repeated measure with an unstructured covariance matrix based on the missing at random assumption; Test type: Other; p = 0.0033, Mixed Models Analysis — Reported p-values are nominal; Least Squares (LS) Mean Difference = -2.3, 95% CI 2-sided [-3.8 to -0.8]

18. Secondary Outcome: Change From Baseline in the European EORTC QLQ HCC 18 Index Score at Cycle 6
Description: The EORTC QLQ-HCC18 is a questionnaire specifically designed to assess health-related quality of life in participants with hepatocellular carcinoma. It includes six symptom scales measuring Fatigue (3 items), Jaundice (2 items), Body Image (2 items), Nutrition (5 items), Pain (2 items), Fever (2 items) and two single items measuring Sex Life and Abdominal Swelling. Participants respond on a scale from 1 = "Not at all" to 4 = "Very Much. Raw scores are transformed into a 0 to 100 scale using linear transformation. The HCC18 Index score is calculated from each of the 6 symptom scales and the 2 single items, and ranges from 0 to 100. Higher scores indicate greater symptom burden or worse quality of life.
  The HEORTC QLQ-HCC18 was not assessed in participants in the sub-study.
Time Frame: Baseline to Cycle 6 (Each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both baseline and Cycle 6 are included
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 166 | 138
score on a scale | 2.2 [0.6 to 3.7] | 4.9 [3.2 to 6.5]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.0096, Mixed Models Analysis — Reported p-values are nominal; LS Mean Difference = -2.7, 95% CI 2-sided [-4.7 to -0.7]

19. Secondary Outcome: Change From Baseline in the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status/Quality of Life Score at Cycle 4
Description: The EORTC QLQ-C30 v3.0 is a questionnaire that assesses quality of life of participants with cancer. It includes global health status and quality of life questions related to overall health in which participants respond based on a 7-point scale, where 1 is very poor and 7 is excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. A higher score indicates better health outcomes.
  The EORTC QLQ-C30 was not assessed in participants in the sub-study.
Time Frame: Baseline to Cycle 4 (each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both Baseline and Cycle 4 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 220 | 176
score on a scale | -0.7 [-3.0 to 1.6] | -5.1 [-7.6 to -2.6]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.0037, Mixed Models Analysis — Reported p-values are nominal; LS Mean Difference = 4.3, 95% CI 2-sided [1.4 to 7.3]

20. Secondary Outcome: Change From Baseline in the EORTC QLQ-C30 Global Health Status/Quality of Life Score at Cycle 6
Description: as for outcome 19
Time Frame: Baseline to Cycle 6 (each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both Baseline and Cycle 6 are included.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 165 | 137
score on a scale | -0.9 [-3.4 to 1.6] | -5.9 [-8.6 to -3.2]
Statistical Analysis 1: Comparison: Arm A: Tislelizumab vs Arm B: Sorafenib; [analysis description as in outcome 17, analysis 1]; Test type: Other; p = 0.0022, Mixed Models Analysis — Reported p-values are nominal; LS Mean Difference = 5.0, 95% CI 2-sided [1.8 to 8.2]

21. Secondary Outcome: Change From Baseline in the European Quality of Life 5 Dimensions, 5-level (EQ-5D-5L) Visual Analogue Scale (VAS) at Cycle 4
Description: The EQ-5D-5L comprises a descriptive module and a Visual Analogue scale (VAS). The EQ-5D-5L VAS measures respondent's self-rated health status on a 0 to 100 scale, with 100 = 'the best health you can imagine' and 0 = 'the worst health you can imagine'. Higher scores on VAS indicate higher health status.
  The EQ-5D-5L VAS was not assessed in participants in the sub-study.
Time Frame: Baseline to Cycle 4 (each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both Baseline and Cycle 4 are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 213 | 170
score on a scale | -0.4 (14.52) | -4.3 (12.92)

22. Secondary Outcome: Change From Baseline in the EQ-5D-5L VAS at Cycle 6
Description: as for outcome 21
Time Frame: Baseline to Cycle 6 (each cycle was 21 days)
Population: ITT Analysis Set. Only participants with data at both Baseline and Cycle 6 are included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 161 | 132
score on a scale | -0.2 (17.03) | -5.4 (13.09)

23. Secondary Outcome: Main Study: Number of Participants With Treatment-emergent Adverse Events
Description: as for outcome 1
Time Frame: From the first dose to 30 days after the last dose, new anticancer therapy, or the study completion analysis cutoff on December 14th, 2023 (a maximum of 61 months for participants in Arm A and 63 months for participants in Arm B).
Population: The Safety Analysis Set includes all randomized participants who received at least one dose of any study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Tislelizumab | Arm B: Sorafenib
Number analyzed (Participants) | 338 | 324
Participants
  TEAEs | 325 | 324
  SAEs | 104 | 91

24. Secondary Outcome: Safety Run-in Sub-study: Number of Participants Who Developed Anti-tislelizumab Antibodies
Description: Treatment-emergent anti-drug antibodies (ADA): participants who were ADA negative at baseline and ADA positive post-baseline.
  Treatment-boosted ADA: participants who were ADA positive at baseline that was boosted to a 4-fold or higher-level following drug administration.
  ADA assessments were not performed for participants enrolled in the main study.
Time Frame: as for outcome 1
Population: The Sub-study Antidrug antibody (ADA) Analysis Set includes all participants enrolled in the sub-study who received at least one dose of tislelizumab for whom both baseline ADA and at least one postbaseline ADA results were available.
Measure: Count of Participants; unit: Participants
Arm/Group | Safety Run-In Sub-study
Number analyzed (Participants) | 10
Participants
  Treatment-Emergent ADA | 1
  Treatment-Boosted ADA | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from informed consent signing to first dose or discontinuation (Screening Period, 28 days) / from first dose to study completion (sub-study, Arm A and Arm B), up to approximately 65 months. AEs are reported from informed consent signing (SAEs only, in the Screening Period; 28 days) / from first dose of study drug to 30 days after last dose, new anticancer therapy, or study completion (up to 64 months in the sub-study, 61 months in Arm A, and 63 months in Arm B).
Description: Results for the sub-study, Arm A, and Arm B are reported for all participants who received treatment (Safety Analysis Set). The Screening Period group includes all enrolled participants, including those who did not receive any study treatment.
  Other (non-serious) adverse events were not collected during the screening period or for participants who did not receive any study treatment.
Groups:
- Screening Period: All Enrolled Participants: All enrolled participants. This group includes deaths and serious adverse events collected from the date of signing the informed consent form and prior to first dose of study drug for participants who received study drug or until study discontinuation for participants who discontinued the study without receiving any study drug.
Arm/Group | Safety Run-In Sub-study | Arm A: Tislelizumab | Arm B: Sorafenib | Screening Period: All Enrolled Participants
All-Cause Mortality (participants affected / at risk) | 7/10 | 258/338 | 273/324 | 1/684
Serious Adverse Events (participants affected / at risk) | 1/10 | 104/338 | 91/324 | 7/684
Other Adverse Events (participants affected / at risk) | 8/10 | 313/338 | 318/324 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In Sub-study (N=10) | Arm A: Tislelizumab (N=338) | Arm B: Sorafenib (N=324) | Screening Period: All Enrolled Participants (N=684)
Cold type haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypersplenism (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Microvascular coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (5) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Anorectal varices (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 4 (4) | 4 (4) | 0 (0)
Chronic gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastric haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Haemoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Intra-abdominal fluid collection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (5) | 1 (1) | 0 (0)
Varices oesophageal (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 0 (0) | 1 (1) | 4 (4) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 3 (3) | 5 (5) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary obstruction (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatic cirrhosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 4 (4) | 3 (3) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hepatic haemorrhage (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Jaundice (Hepatobiliary disorders) | 0 (0) | 3 (3) | 5 (5) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Jaundice hepatocellular (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 5 (5) | 3 (3) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hepatic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Radiation oesophagitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 5 (5) | 4 (4) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 6 (7) | 5 (5) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Hepatic enzyme abnormal (Investigations) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (5) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumour rupture (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiplegia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic fluid collection (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Hepatopulmonary syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pulmonary alveolar haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Acute generalised exanthematous pustulosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Immune-mediated dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Radiotherapy (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Shock haemorrhagic (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Run-In Sub-study (N=10) | Arm A: Tislelizumab (N=338) | Arm B: Sorafenib (N=324) | Screening Period: All Enrolled Participants (N=0)
Anaemia (Blood and lymphatic system disorders) | 3 (3) | 41 (73) | 32 (47) | NA
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 14 (29) | 18 (26) | NA
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 3 (21) | 13 (16) | NA
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 15 (24) | 31 (47) | NA
Palpitations (Cardiac disorders) | 1 (2) | 2 (2) | 4 (4) | NA
Vertigo (Ear and labyrinth disorders) | 1 (2) | 5 (5) | 1 (1) | NA
Hyperthyroidism (Endocrine disorders) | 0 (0) | 15 (15) | 4 (4) | NA
Hypothyroidism (Endocrine disorders) | 0 (0) | 29 (33) | 12 (12) | NA
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 32 (36) | 20 (25) | NA
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 38 (47) | 40 (51) | NA
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 18 (20) | 32 (40) | NA
Ascites (Gastrointestinal disorders) | 0 (0) | 14 (14) | 8 (8) | NA
Constipation (Gastrointestinal disorders) | 0 (0) | 28 (35) | 28 (36) | NA
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 38 (52) | 142 (379) | NA
Dry mouth (Gastrointestinal disorders) | 0 (0) | 11 (13) | 10 (11) | NA
Dyspepsia (Gastrointestinal disorders) | 1 (2) | 14 (15) | 10 (18) | NA
Nausea (Gastrointestinal disorders) | 0 (0) | 27 (29) | 33 (34) | NA
Stomatitis (Gastrointestinal disorders) | 1 (2) | 9 (10) | 17 (23) | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 25 (31) | 16 (25) | NA
Asthenia (General disorders) | 0 (0) | 34 (40) | 26 (34) | NA
Fatigue (General disorders) | 3 (3) | 36 (40) | 37 (48) | NA
Infusion site extravasation (General disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Malaise (General disorders) | 0 (0) | 13 (13) | 14 (15) | NA
Oedema peripheral (General disorders) | 2 (2) | 21 (25) | 16 (16) | NA
Pyrexia (General disorders) | 4 (4) | 56 (77) | 56 (75) | NA
Hepatic pain (Hepatobiliary disorders) | 0 (0) | 13 (16) | 12 (14) | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 14 (25) | 16 (30) | NA
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 1 (1) | 0 (0) | NA
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | NA
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | NA
Herpes zoster (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | NA
Influenza (Infections and infestations) | 1 (1) | 5 (5) | 2 (2) | NA
Nasopharyngitis (Infections and infestations) | 2 (2) | 11 (13) | 11 (13) | NA
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 4 (4) | NA
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | NA
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 30 (40) | 13 (15) | NA
Urinary tract infection (Infections and infestations) | 1 (2) | 12 (13) | 12 (15) | NA
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) | NA
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | NA
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 1 (1) | NA
Alanine aminotransferase increased (Investigations) | 0 (0) | 93 (133) | 111 (168) | NA
Amylase increased (Investigations) | 1 (1) | 0 (0) | 4 (5) | NA
Aspartate aminotransferase increased (Investigations) | 1 (1) | 124 (179) | 135 (213) | NA
Bilirubin conjugated increased (Investigations) | 0 (0) | 28 (40) | 33 (56) | NA
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 42 (69) | 37 (52) | NA
Blood bilirubin increased (Investigations) | 1 (1) | 74 (143) | 101 (167) | NA
Blood bilirubin unconjugated increased (Investigations) | 0 (0) | 12 (19) | 13 (25) | NA
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 17 (20) | 13 (17) | NA
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 20 (27) | 13 (26) | NA
Blood creatinine increased (Investigations) | 1 (1) | 9 (17) | 3 (5) | NA
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 24 (33) | 28 (55) | NA
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 43 (61) | 42 (51) | NA
Hepatitis C RNA increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | NA
Neutrophil count decreased (Investigations) | 1 (1) | 30 (65) | 29 (59) | NA
Platelet count decreased (Investigations) | 0 (0) | 50 (81) | 69 (106) | NA
Weight decreased (Investigations) | 0 (0) | 35 (40) | 63 (72) | NA
White blood cell count decreased (Investigations) | 0 (0) | 32 (63) | 31 (69) | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 45 (53) | 57 (60) | NA
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 2 (2) | 0 (0) | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 19 (54) | 18 (24) | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 45 (81) | 32 (44) | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 7 (9) | 15 (22) | NA
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 21 (43) | 34 (63) | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (24) | 12 (18) | NA
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 20 (26) | 28 (34) | NA
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 9 (21) | 45 (78) | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 (0) | 9 (12) | 10 (12) | NA
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 40 (54) | 22 (30) | NA
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 29 (32) | 20 (24) | NA
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (6) | 12 (16) | NA
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 11 (17) | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 11 (11) | 12 (18) | NA
Dizziness (Nervous system disorders) | 1 (1) | 12 (16) | 8 (10) | NA
Dysgeusia (Nervous system disorders) | 1 (1) | 5 (6) | 2 (2) | NA
Headache (Nervous system disorders) | 0 (0) | 16 (19) | 17 (20) | NA
Insomnia (Psychiatric disorders) | 1 (1) | 19 (20) | 17 (21) | NA
Proteinuria (Renal and urinary disorders) | 0 (0) | 11 (15) | 12 (12) | NA
Renal impairment (Renal and urinary disorders) | 1 (1) | 1 (1) | 1 (1) | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 38 (44) | 25 (27) | NA
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 28 (30) | NA
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 12 (13) | 8 (8) | NA
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (5) | 8 (10) | NA
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 5 (6) | 12 (15) | NA
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 75 (76) | NA
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (5) | 1 (1) | NA
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 12 (13) | 6 (7) | NA
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 11 (11) | NA
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (4) | 0 (0) | NA
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 203 (231) | NA
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 48 (58) | 25 (28) | NA
Rash (Skin and subcutaneous tissue disorders) | 3 (4) | 40 (50) | 56 (65) | NA
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 4 (4) | 15 (17) | NA
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | NA
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 1 (2) | NA
Hypertension (Vascular disorders) | 1 (3) | 23 (27) | 90 (126) | NA
Hypotension (Vascular disorders) | 1 (1) | 5 (5) | 2 (2) | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period,Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (3):
  • Study Protocol (2020-05-11): https://cdn.clinicaltrials.gov/large-docs/73/NCT03412773/Prot_000.pdf
  • Statistical Analysis Plan: SAP for Primary Analysis CSR (2022-04-21): https://cdn.clinicaltrials.gov/large-docs/73/NCT03412773/SAP_001.pdf
  • Statistical Analysis Plan: SAP for Study Closeout Analysis CSR (2023-12-22): https://cdn.clinicaltrials.gov/large-docs/73/NCT03412773/SAP_002.pdf